CLINICAL TRIAL: NCT07301710
Title: Myofunctional Therapy for Obstructive Sleep Apnea in U.S. Service Members With and Without Traumatic Brain Injury
Brief Title: Low-Tech Treatments for Obstructive Sleep Apnea
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WRNMMC-2025-0481; US240046 (Other Grant/Funding Number: Uniformed Services University of the Health Sciences)
Record Dates: First submitted 2025-11-05; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea (OSA); Traumatic Brain Injury (TBI)
Keywords: Obstructive Sleep Apnea; Myofunctional Therapy; Traumatic Brain Injury; Randomized Controlled Trial; Oropharyngeal Exercises; Respiratory Resistance Training
MeSH Terms: conditions — Sleep Apnea, Obstructive; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofunctional Therapy (Experimental)
  Interventions: Behavioral: High-Resistance Breathing and Drinking Exercises
- Relaxation Therapy (Sham Comparator)
  Interventions: Behavioral: Low-Resistance Breathing and Drinking Exercises

INTERVENTIONS:
Behavioral: High-Resistance Breathing and Drinking Exercises — Three months of drinking at least 32-oz of water daily through a high-resistance nozzle, and inhaling and exhaling 60 times per day through a high-resistance breathing device
  Other Names: Device-Assisted Myofunctional Therapy
  Arms: Myofunctional Therapy
Behavioral: Low-Resistance Breathing and Drinking Exercises — Three months of drinking 32-oz of water daily through a low-resistance nozzle, and inhaling and exhaling 60 times per day through a low-resistance breathing device
  Other Names: Placebo Therapy
  Arms: Relaxation Therapy

SUMMARY:
The overall purpose of this study is to compare changes in sleep outcomes in people with obstructive sleep apnea (OSA) depending on their participation in one of two behavioral interventions; both involve drinking water and breathing. A second purpose is to compare outcomes between people who have sustained a traumatic brain injury (TBI) and those with no history of TBI. The main questions it aims to answer are whether sleep quality improves after 3-months of high-resistance versus low-resistance exercises, and whether people have different outcomes depending on their history of TBI.

DETAILED DESCRIPTION:
Background

A nonintrusive, inexpensive behavioral approach is emerging as a promising alternative to the management of obstructive sleep apnea (OSA). Generally referred to as myofunctional therapy (MFT), the approach involves exercising the muscles of the oropharynx and respiratory system.The exercises are intended to improve muscle strength and tone so that the muscular structures of the upper airway improve their neuromuscular responsiveness to breathing and resist collapsing into the airway during sleep. They are relatively simple to implement and train, but the regimen requires high-dosage practice and strict dedication to habituate. There is a need for an MFT protocol to be delivered in a consistent manner that is simple, sustainable, and motivating. This study takes advantage of recent low-tech tools that appear to elicit the desired muscle actions achieved with MFT.

Participant Recruitment

Participants are recruited from the Sleep Clinic at Walter Reed National Military Medical Center if they receive a new diagnosis of obstructive sleep apnea (AHI >5) based on standard-of-care polysomnography (PSG) or if they do not successfully use a standard first-line treatment. After providing informed consent and passing screening tests, they are randomized into one of two behavioral interventions.

Interviews will determine whether participants have a history of TBI. Participants in the two intervention arms will be block stratified based on +/- TBI and TBI severity. The groups will also be stratified based on OSA severity.

Interventions

The interventions involving drinking water through a study-provided water bottle with a specially designed nozzle and breathing in and out through a study-provided handheld breathing device multiple times daily for 3 months. Therefore, this novel intervention is called "HydroBreathe Therapy." The intervention arms are named for the color of the breathing device. Participants will be informed that the Green option involves exercises intended to relax airway structures and promote better airway patency, and that the Black option involves high-resistance exercises intended to increase airway muscle strength to resist structural collapse. Participants are not informed which of the options is expected to be more therapeutic, but they are informed that both may help and neither will worsen their OSA.

Participants will enter their daily practice into electronic adherence logs, which will be monitored by the study team. A study team member will contacted participants every 2 weeks throughout the intervention period to offer encouragement and answer questions.

Assessments

Pre- and post-intervention measures are obtained from PSG results, self-assessment questionnaires, and measures of tongue and respiratory muscle function. Participants in the experimental group will be given the option to participate in a 3-week follow-up assessment including the questionnaires and muscle-function testing if they are willing to delay first-line treatment for OSA. All participants will be referred back to the Sleep Clinic for standard treatment at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of OSA (AHI, ≥ 5) or failure of first-line OSA treatment;
* Willingness to forego first-line OSA treatment or stop current OSA treatment for 3 months;
* Ability to follow directions and perform the required exercises;
* Age between 18-65 yr.

Exclusion Criteria:

* Current use of OSA treatment;
* Medical comorbidities that require restricting fluid intake (e.g., dysphagia, renal disease, liver disease, hyponatremia);
* Severe nasal obstruction; 4) severe ankyloglossia; 4) craniofacial abnormality; 5) severe pulmonary disease; 6) severe post-traumatic stress disorder; 7) very severe insomnia; 8) body mass index (BMI) ≥30 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | From enrollment to end of three-month intervention
  AHI is the number of apneic and hypopneic episodes per hour of sleep. The scores start at zero, meaning no events are taking place. A mild score falls in the range of 5-15; moderate 15-30, and a severe diagnosis is 30 or more events per hour. Pre-intervention AHI is obtained from standard-of-care in-clinic sleep study. Post-intervention AHI is obtained from an in-clinic sleep study conducted as part of this research.

SECONDARY OUTCOMES:
SpO2 | From enrollment to end of three-month intervention
  Oxygen saturation measured during the in-clinic sleep studies. Normal levels range between 95-100%.
Snore Index | From enrollment to end of three-month intervention
  Number of snoring episodes per hour of sleep
Epworth Sleepiness Scale (ESS) | From enrollment to end of three-month intervention with option for additional three-week follow-up
  A self-assessment of daytime sleepiness
Functional Outcomes of Sleep Questionnaire-10 (FOSQ-10) | From enrollment to end of three-month intervention with option for additional three-week follow-up
  A self-assessment of impact of daytime sleepiness

OTHER OUTCOMES:
Tongue Strength | From enrollment to end of three-month intervention with option for additional three-week follow-up
  The maximum pressure generated during tongue-to-palate compression of an air-filled bulb over three trials
Tongue Endurance | From enrollment to end of three-month intervention with option for additional three-week follow-up
  The maximum duration of sustaining tongue-to-palate compression of an air-filled bulb at 50% of maximum pressure.
Maximal Inspiratory Pressure (MIP) | From enrollment to end of three-month intervention with option for additional three-week follow-up
  The maximum pressures generated during maximal-effort inspiration in cmH2O.
Maximal Expiratory Pressure (MEP) | From enrollment to end of three-month intervention with option for additional three-week follow-up
  The maximum pressures generated during maximal-effort expiration in cmH2O.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes